CLINICAL TRIAL: NCT02355951
Title: Non-investigational Study to Evaluate Adenovirus Serotype 5 (Ad5) Neutralizing Antibodies (nAb) in Patients With Chronic Hepatitis B Virus (HBV) Mono-infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: TG1050.01
Record Dates: First submitted 2015-01-21; First posted 2015-02-04 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood draw

SUMMARY:
Objectives:

Primary Objective:

To identify and preselect patients with chronic HBV mono infection, who are undetectable for anti-Ad5 nAb, currently being treated with nucleo(t)sides, for participation in the TG1050.02 Phase1/1b First in Man (FIM) study.

Secondary Objectives:

To assess the prevalence of undetectable anti-Ad5 nAb in chronic HBV mono-infected patients.

Methodology:

Patients with chronic HBV mono-infection, who are currently being treated with nucleo(t)sides for their HBV infection, will be enrolled in this study to measure Ad5 nAb levels. A single peripheral blood collection (4 mL) will be obtained and Ad5 nAb titers will be measured by a central laboratory using a newly validated assay.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 65 years of age, inclusive
* Patients mono-infected with HBV and currently on HBV treatment for at least 2 years with either the nucleos(t)ide tenofovir (TDF) or entecavir (ENT)
* HBV DNA < lower limit of quantification (LLOQ) (eg, HBV deoxyribonucleic acid (DNA) < 20 IU/mL using the Roche COBAS TaqMan assay) within 6 last months
* Signed, written Independent Ethics Committee (IEC)-approved informed consent

Exclusion Criteria:

* Patients with either medical history or evidence of cirrhosis, as documented in the medical source, who had: a) any biopsy showing cirrhosis; or b) any transient elastography score of ≥ 10.5 kPa or Fibrosure® / FibroTest ® score of ≥ 0.48 with either test result within past 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Immunology analysis: Serum titers of Adenovirus serotypes 5 (Ad5) neutralizing antibodies (nAb) | Day 1

CONTACTS AND LOCATIONS:
Locations (11):
- Montreal, Canada
- France (5):
  - Grenoble
  - Lyon
  - Nancy
  - Paris
  - Strasbourg
- Germany (5):
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Mainz
  - München